CLINICAL TRIAL: NCT00334386
Title: Multicentre, Multinational, Parallel, Randomised, Double Blind Clinical Trial, to Evaluate the Non-inferiority of PR Torasemide Versus IR Torasemide in Patients With Mild or Moderate Arterial Hypertension.
Brief Title: Hypertension Study: Multinational Torasemide Trial in Mild to Moderate Hypertension.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P030089-01; EudraCT: 2004-000876-14
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: Hypertension; Anti-hypertensive effect; Diuretic
MeSH Terms: conditions — Hypertension | interventions — Sodium Potassium Chloride Symporter Inhibitors; Torsemide

INTERVENTIONS:
Drug: Torasemide Prolonged Release (loop diuretic)
Drug: Torasemide Immediate Release (loop diuretic)

SUMMARY:
Primary objective:To demonstrate the no-inferiority in efficacy of treatment with Torsemide-PR in relation to Torsemide-IR in patients with mild and/or moderate hypertension.

Secondary objectives: To evaluate the safety and tolerability of Torsemide-PR.

DETAILED DESCRIPTION:
Torsemide is a loop diuretic from the group of pyridine-sulfonylureas, which acts on the ascending large portion of the Henle loop where it inhibits the Na+/K+/2Cl- transport!system and blocks Cl- channels.Therefore, sodium and chlorine ions and water can not be reabsorbed in the tubule and the urine volume increases significantly. Torsemide is used for the treatment of oedema associated with congestive heart failure, kidney or liver disease and, either alone or combined with other anti-hypertensive drugs, for the treatment of arterial hypertension.

This trial compares the effect of a new formulation of Torasemide (Torasemide prolonged release)to the already available immediate release formulation of the same drug on the treatment of mild to moderate hypertensive patients.

Eligible patients will be randomised to either treatment with Torasemide prolonged release or with Torasemide immediate release and will be followed-up until completing 3 months of treatment.Blood pressure will be measured by an OMRON pressure gauge. Additionally, ABPM will be performed on a sub-group of the patients taking part in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 75, inclusive.
2. Ambulatory patients diagnosed with mild or moderate arterial hypertension complying with the following requirements:

   1. Patients diagnosed "de novo".
   2. Patients with prior anti-hypertensive treatment in monotherapy who do not respond to the treatment and, in the investigator's opinion, could benefit from diuretic treatment in monotherapy.
   3. Patients with prior anti-hypertensive treatment in monotherapy who do not tolerate the current treatment and, in the investigator's opinion, could benefit from diuretic treatment in monotherapy.

   Patients with prior treatment must be able to interrupt their present treatment for a period of up to 3 months.

   (Mild or moderate hypertension defined by blood pressure levels: Systolic blood pressure from 140-179 mm Hg and diastolic blood pressure from 90-109 mm Hg) (2003 European Society of Hypertension-European Society of Cardiology guidelines for management of arterial hypertension) (3)
3. Capable of understanding the nature of the trial.
4. Providing their informed consent in writing.

Exclusion Criteria:

1. Pregnant or breastfeeding women and women of fertile age who are not using a safe contraceptive method or do not intend to use one during the trial. Safe contraceptive methods are oral or parenteral contraceptive treatments or barrier methods: masculine or feminine condom, diaphragm and/or IUD.
2. Severe arterial hypertension (systolic blood pressure of 180 mmHg or above and diastolic blood pressure of 110 mmHg or above).
3. Known or suspected secondary arterial hypertension.
4. History of known hypersensitivity to the compound under study or to sulfonylureas.
5. History of repeated and documented hypertensive crises.
6. NYHA grade II to IV congestive heart failure.
7. Severe cardiac arrhythmia (sustained ventricular tachycardia, auricular fibrillation, auricular flutter, bradycardia under 45 beats per minute).
8. Unstable angina pectoris.
9. Acute myocardial infarct in the last 6 months.
10. Liver failure defined by the following analytical parameters: - SGPT (ALT) or SGOT (AST) over twice the upper normal limit.
11. Chronic kidney failure defined by the following analytical parameters: Serum creatinine over 2.3 mg/dl (or 203 mol/L).
12. Patients with insulin-dependent diabetes and patients with non-insulin dependent diabetes.
13. Cerebrovascular accident in the last 6 months.
14. Contraindications in the data obtained during the selection process in the physical examination, haematology, biochemistry, urine analysis and 12-lead ECG, in the investigator's opinion.
15. Simultaneous participation in another clinical trial or treatment with any investigational drug within the 30 days prior to signing the informed consent form.
16. Lactose intolerance.
17. Concomitant treatment with lithium.
18. Patients requiring chronic treatment (treatment > 7 days) with non-steroidal anti-inflammatory drugs, including aspirin.
19. Patients with concomitant treatment with aminoglycoside antibiotics, etacrynic acid.
20. Chronic administration of any medication affecting blood pressure.
21. Patients in treatment with group 1a, 1b or 2 anti-arrhythmic drugs.
22. History of drug or alcohol addiction within the 6 months prior to the start of the trial.
23. Any clinical circumstance or condition which, in the investigator's opinion, could affect the possibility of completing the protocol and the administration of Torasemide.
24. Obesity with a body mass index (BMI) of over 40 kg/m2.
25. Patients who do not respond to diuretic treatment in monotherapy.
26. Patients with prior anti-hypertensive treatment in monotherapy who are candidates for anti-hypertensive treatment in polytherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388
Dates: Start 2005-04; Study Completion 2006-02

PRIMARY OUTCOMES:
Difference in mm Hg between the mean diastolic blood pressure (DBP) values the baseline period and the values at the end of the treatment period.

SECONDARY OUTCOMES:
Difference in mm Hg, systolic blood pressure (SBP) values in the baseline period and the values at the end of the treatment period.
Percentage of patients with controlled blood pressure (SBP < 140 and/or DBP < 90) at the end of the treatment period.
Urinary symptoms.
ABPM values measured in a subgroup of patients
Safety & tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Roca, MD, PhD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Antonio Coca, MD, PhD, Principal Investigator — H. Clínic Barcelona, Barcelona, Spain; Joaquim Vila, MD, Principal Investigator — Hospital Municipal de Badalona, Badalona, Barcelona, Spain; Javier Sobrino, MD, Principal Investigator — Hospital del Esperit Sant, Santa Coloma de Gramanet, Barcelona, Spain; Jaume Plana, MD, Principal Investigator — Hospital Residencia Sant Camil, Sant Pere de Ribes, Barcelona, Spain; Xavier Farres, MD, Principal Investigator — Centre d'Atenció Primaria El Remei de Vic, Vic, Barcelona, Spain; Joan Garcia, MD, PhD, Principal Investigator — Hospital Universitario La Paz; Manuel Luque, MD, Principal Investigator — Hospital Clínico San Carlos, Madrid, Spain; Luis De Teresa, MD, Principal Investigator — Hospital de Sant Vicenç de Raspeig, Sant Vicenç de Raspeig, Alicante, Spain; Jose Vicente, MD, Principal Investigator — Centro de Salud de Petrel, Petrel, Alicante, Spain; Angela Felip, MD, PhD, Principal Investigator — Hospital de Mataró, Mataró, Barcelona, Spain; Pedro Aranda, MD, PhD, Principal Investigator — Hospital Universitario Carlos Haya, Málaga, Spain; Pablo Gómez, MD, PhD, Principal Investigator — Hospital de Jerez de la Frontera, Cádiz, Spain; Blas Gil, MD, Principal Investigator — Hospital Clínico Universitario San Cecilio, Granada, Spain; Joaquín Aracil, MD, Principal Investigator — Centro de Salud El Cristo, Oviedo, Asturias, Spain; Miguel A Prieto, MD, Principal Investigator — Centro de Salud Vallobin Concinos, Oviedo, Asturias, Spain; Carles Brotons, MD, PhD, Principal Investigator — Centre d'Atenció Primaria Sardenya, Barcelona, Spain; Félix Laporta, MD, Principal Investigator — Centro de Salud La Roda, La Roda, Albacete, Spain; José A División, MD, Principal Investigator — Centro de Salud de Fuentealbilla, Fuentealbilla, Albacete, Spain; Enrique López, MD, Principal Investigator — Centro de Salud de Chinchilla, Chinchilla, Albacete, Spain; Carlos Calvo, MD, PhD, Principal Investigator — Hospital Universitario de Santiago, Santiago de Compostela, Spain; Emili Marco, MD, Principal Investigator — Centre d'Atenció Primaria de Sarrià de Ter, Sarrià de Ter, Girona, Spain; Joan Martorell, MD, Principal Investigator — Centre de Salut de Guisona, Guisona, Lleida, Spain; Montserrat Pujol, MD, Principal Investigator — Centre d'Atenció Primaria El Carmel, Barcelona, Spain; Raquel Adroer, MD, Principal Investigator — Centre d'Atenció Primaria Florida Nord, Barcelona, Spain; Angel Cano, MD, Principal Investigator — Centre d'Atenció Primaria Bon Pastor, Barcelona, Spain; Nadezhda S Alexeeva, PhD, Principal Investigator — St. Petersburg Cardiology Clinic, St. Petesburg, Russia; Andrei Y Baranovsky, MD, PhD, Principal Investigator — St. Petersburg City Hospital #31, St. Petesburg, Russia; Svetlana A Boldueva, MD, PhD, Principal Investigator — St. Petersburg Mechnikov State Medical Academy, St. Petesburg, Russia; Svetlana K Churina, MD, PhD, Principal Investigator — Pokrovskaya Hospital, 1-st and 2-nd Cardiology Department, St. Petesburg, Russia; Boris M Goloschekin, MD, PhD, Principal Investigator — St. Petersburg City Hospital #15, St. Petesburg, Russia; Yanis Y Dumpis, MD, Principal Investigator — St.Petersburg Mechnikov State Medical Academy North-West Center of Arrhythmia Diagnostics and Treatment, St. Petesburg, Russia; Konstantin N Zrazhevsky, MD, PhD, Principal Investigator — St.Petersburg City Hospital #8, St. Petesburg, Russia; Victor Kostenko, MD, PhD, Principal Investigator — St.Petersburg City Outpatient Unit #109, St. Petesburg, Russia; Elena F Pavlysh, MD, PhD, Principal Investigator — St.Petersburg City Outpatient Unit #25, St. Petesburg, Russia; Lev A Sorokin, MD, PhD, Principal Investigator — St. Elizabeth City Hospital, St. Petesburg, Russia; Irina A Zobenko, MD, Principal Investigator — JSC Chernaya Rechka Health Center, St. Petesburg, Russia; Alexander O Sherenkov, MD, PhD, Principal Investigator — Krasnogvardeysky District Medical-Physiology Clinic, St. Petesburg, Russia; Alexander V Orlov-Morozov, MD, PhD, Principal Investigator — Moscow City Hospital #23, Moscow, Russia; Vladimir A Parfenov, MD, PhD, Principal Investigator — Moscow City Hospital #61, Moscow, Russia; Victor A Milyagin, MD, PhD, Principal Investigator — Smolensk State Medical Academy, Smolensk, Russia